CLINICAL TRIAL: NCT01754389
Title: A 3-Arm Randomized Phase II Study of Standard-of-Care vs. Bortezomib Based Graft-Versus-Host Disease Regimen for Reduced-Intensity Conditioning Hematopoietic Stem Cell Transplantation Patients Lacking HLA-matched Related Donors
Brief Title: Standard of Care vs. Bortezomib in Graft-Versus Host Disease After Hematopoietic Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, John Koreth, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-404
Record Dates: First submitted 2012-12-13; First posted 2012-12-21 (Estimated); Results first posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-06

CONDITIONS: Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Tacrolimus; Methotrexate; Bortezomib; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (Standard of Care) (Active Comparator): Tacrolimus intravenously and orally, Day -3 through 3-6 months post-transplant Methotrexate intravenously on days 1, 3, 6 and 11 post-transplant
  Interventions: Drug: Tacrolimus; Drug: Methotrexate
- Arm B (Experimental) (Experimental): Bortezomib intravenously 1, 4 and 7 days post-transplant Tacrolimus intravenously and orally, Day -3 through 3-6 months post-transplant Methotrexate intravenously 1,3,6 and 11 days post-transplant
  Interventions: Drug: Tacrolimus; Drug: Methotrexate; Drug: Bortezomib
- Arm C (Experimental) (Experimental): Bortezomib intravenously 1,4 and 7 days post-transplant Sirolimus, intravenously and orally, Day -3 through 3-6 months post-transplant Tacrolimus, intravenously and orally, Day -3 through 3-6 months post-transplant
  Interventions: Drug: Tacrolimus; Drug: Bortezomib; Drug: Sirolimus

INTERVENTIONS:
Drug: Tacrolimus
Drug: Methotrexate
  Arms: Arm A (Standard of Care); Arm B (Experimental)
Drug: Bortezomib
  Arms: Arm B (Experimental); Arm C (Experimental)
Drug: Sirolimus
  Arms: Arm C (Experimental)

SUMMARY:
This research study is a Phase II clinical trial. Phase II clinical trials test the effectiveness of an investigational drug to learn whether the drug works in treating a specific cancer. "Investigational" means that the drug is still being studied and that research doctors are trying to find out more about it-such as the safest dose to use, the side effects it may cause, and if the drug is effective for treating different types of cancer. It also means that the FDA has not yet approved bortezomib to treat or prevent graft-versus-host disease. Bortezomib is approved by the FDA to treat other human malignancies.

Bortezomib is a drug that has an anti-cancer effect that involves inhibiting cell growth and causing cell death. This drug has been used in other research studies, and information from thos other research studies suggests that bortezomib may help to lower the risk of GVHD after allogeneic stem cell transplantation in patients who have matched unrelated, unmatched related or unrelated donors in this research study.

Allogeneic stem cell transplantation is a procedure in which selected blood cells taken from your sibling or unrelated donor are given to you. Lower doses of chemotherapy drugs are given before the donor cells are infused in a process known as reduced-intensity conditioning. Stem cell transplant destroys cancer in two ways: The conditioning regimen destroys cancer cells and teh immune cells from the donor can recognize cancer cells and kill them.

A common problem after stem cell transplant is graft-versus-host disease (GVHD). The word "graft" refers to the donor blood cells that you will receive during your transplant. The word "host" refers to the person (in this case, you) receiving the cells. GVHD is a complication of transplantation where the donor graft attacks and damages some of your tissues. GVHD can cause skin rash, intestinal problems such as nausea, vomiting or diarrhea. GVHD may also damage your liver and cause hepatitis or jaundice. GVHD may also increase your risk of infection.

After stem cell transplant, all patients receive prophylactic medications against GVHD. In this research study we are studying the safety and effectiveness of preventing GVHD using bortezomib treatment in combination with other drugs versus standard of care prophylaxis (tacrolimus + methotrexate). If you take part in this study, there is a 33% chance you will receive any one of the following GVHD prevention treatments:

* tacrolimus + methotrexate (standard of care GVHD prophylaxis)
* bortezomib + tacrolimus + methotrexate
* bortezomib + sirolimus + tacrolimus Sirolimus, tacrolimus and methotrexate are drugs that suppress the immune system to try to prevent GVHD.

DETAILED DESCRIPTION:
You will undergo some screening tests or procedures to find out if you can be in this research study. Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out that you do not take part in the research study. If you have had some of these tests or procedures recently, they may or may not have to be repeated. Possible tests include a medical history, physical exam, laboratory tests, pulmonary function tests, cardiac ejection fraction and a pregnancy test. If these tests show that you are eligible to participate in the research study, you will begin the study treatment. If you do not meet the eligibility criteria, you will not be able to participate in the research study.

Because no one knows which of the study options is best, you will be "randomized" into one of the study groups (described below). Randomization means that you are put into a group by chance. It is like flipping a coin. You will have an equal chance of being placed in any of the groups.

Before your transplant you will receiving conditioning therapy. The conditioning therapy for this study involves fludarabine and busulfex. These drugs will be given five, four, three and two days before your transplant (Days -5 through -2). Both these chemotherapy drugs are commonly used in allogeneic stem cell transplantation. On Day 0, you will receive selected blood cells taken from your sibling or unrelated donor.

You will receive 1 of 3 GVHD prophylaxis plans depending on which one you are randomized to:

* Arm A will receive tacrolimus + methotrexate
* Arm B will receive bortezomib + tacrolimus + methotrexate
* Arm C will receive bortezomib + sirolimus + tacrolimus

Tacrolimus (Arm A, B and C) will be started three days before your transplant (Day -3). You will be given tacrolimus initially intravenously (through a needle in a vein in your arm or through a "central line", a catheter or tube placed in the large vein under your collarbone or your neck) and later by mouth. You will continue to take tacrolimus for 3 to 6 months after your transplant. Your physician will discuss your tacrolimus dose with you.

Methotrexate (Arms A and B) will be given intravenously one, three, six and eleven days after your transplant (Days 1,3,6 and 11).

Bortezomib (Arms B and C) will be given intravenously one, four and seven days after your transplant (Days 1,4 and 7).

Sirolimus (Arm C only) will start three days before your transplant (Day -3). You will be given sirolimus initially intravenously and then later by mouth. You will need to continue to take your sirolimus for 3 to 6 months after your transplant. Your physician will discuss your sirolimus dose with you.

To help with engraftment, you will be given the drug G-CSF (Neupogen) starting the day after your transplant, until your white blood cells recover. You will receive other medications as part of standard of care to help prevent you from getting infections. You will also receive medications to help prevent seizures during your conditioning therapy.

Each week for the first four weeks and 2,3,6 and 12 months following your transplant, you will have a physical exam and you will be asked questions about your general health and specific questions about any problems that you might be having and any medications you may be taking. If you are taking bortezomib, you will have an exam and may be asked to fill out an additional questionnaire about potential symptoms of numbness, tingling, weakness or pain on days 1,4 and 7 after your transplant.

Each week for the first four weeks and 12 months following your transplant, you will have blood drawn (approximately 6 teaspoons) to monitor your progress and health following transplant. If you receive methotrexate and/or bortezomib, you will have an additional blood draw on those days.

Approximately 12 months following your transplant, a needle will be inserted into your hip bone and a small amount of bone marrow cells and a sample of bone are removed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced/aggressive hematologic malignancy unlikely to be cured by alternative therapies
* HLA matched unrelated donors or 1-locus HLA mismatched related or unrelated donors
* Adequate organ function
* Willing to use appropriate contraception

Exclusion Criteria:

* Pregnant or breastfeeding
* Recipient of prior allogeneic hematopoietic stem cell transplantation
* Recipient of prior abdominal radiation therapy
* HIV positive on combination anti-retroviral therapy
* Seropositive for hepatitis B or C
* Known allergy to bortezomib, boron or mannitol
* Myocardial infarction within 6 months prior to enrollment or any other cardiac dysfunction
* Uncontrolled infection
* Inability to withhold agents that may interact with hepatic cytochrome P450 enzymes or gluthathione S-transferases
* Seizures or history of seizures
* Grade greater than or equal to 2 peripheral neuropathy within 21 days of enrollment
* Use of other investigational drugs within 21 days of enrollment
* History of another non-hematologic malignancy except if disease free for at least 5 years or cervical cancer in situ, or basal/squamous cell carcinoma of the skin
* Uncontrolled intercurrent illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2013-01; Primary Completion 2016-05 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Koreth, DPhil, MBBS, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Insitute, Boston, Massachusetts

REFERENCES:
- [Derived] Koreth J, Kim HT, Lange PB, Poryanda SJ, Reynolds CG, Rai SC, Armand P, Cutler CS, Ho VT, Glotzbecker B, Yusuf R, Nikiforow S, Chen YB, Dey B, McMasters M, Ritz J, Blazar BR, Soiffer RJ, Antin JH, Alyea EP 3rd. Bortezomib-based immunosuppression after reduced-intensity conditioning hematopoietic stem cell transplantation: randomized phase II results. Haematologica. 2018 Mar;103(3):522-530. doi: 10.3324/haematol.2017.176859. Epub 2018 Jan 11. PMID 29326124

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Excluded (n= 4)
  * Not meeting inclusion criteria (n=3;active infection (2*), disease relapse (2*))
  * Declined to participate (n=1; interacting medication per provider preference (1))
Groups:
- Arm A (Standard of Care): Drug: Tacrolimus, Methotrexate
  Tacrolimus intravenously and orally, Day -3 through 3-6 months post-transplant Methotrexate intravenously on days 1, 3, 6 and 11 post-transplant
- Arm B (Experimental): Drug: Bortezomib, Tacrolimus, Methotrexate Other Names: Velcade
  Bortezomib intravenously 1, 4 and 7 days post-transplant Tacrolimus intravenously and orally, Day -3 through 3-6 months post-transplant Methotrexate intravenously 1,3,6 and 11 days post-transplant
- Arm C (Experimental): Drug: Bortezomib, Sirolimus, Tacrolimus Other Names: Velcade
  Bortezomib intravenously 1,4 and 7 days post-transplant Sirolimus, intravenously and orally, Day -3 through 3-6 months post-transplant Tacrolimus, intravenously and orally, Day -3 through 3-6 months post-transplant
Period: Overall Study
Arm/Group | Arm A (Standard of Care) | Arm B (Experimental) | Arm C (Experimental)
Started | 46 | 45 | 47
Completed | 46 | 45 | 47
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm B (Experimental): Drug: Bortezomib, Tacrolimus, Methotrexate Other Names: Velcade
  Bortezomib intravenously 1, 4 and 7 days post-transplant Tacrolimus intravenously and orally, Day -3 through 3-6 months post-transplant Methotrexate intravenously 1,3,6 and 11 days post-transplant
  Bortezomib
- Arm C (Experimental): Drug: Bortezomib, Sirolimus, Tacrolimus Other Names: Velcade
  Bortezomib intravenously 1,4 and 7 days post-transplant Sirolimus, intravenously and orally, Day -3 through 3-6 months post-transplant Tacrolimus, intravenously and orally, Day -3 through 3-6 months post-transplant
  Sirolimus
- Total: Total of all reporting groups
Arm/Group | Arm A (Standard of Care) | Arm B (Experimental) | Arm C (Experimental) | Total
Number analyzed (Participants) | 46 | 45 | 47 | 138
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 22 | 29 | 70
  >=65 years | 27 | 23 | 18 | 68
Age, Continuous [Median (Full Range); unit: years] | 65 [29 to 74] | 65 [30 to 75] | 62 [24 to 73] | 64 [24 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 13 | 23 | 54
  Male | 28 | 32 | 24 | 84
Region of Enrollment [Number; unit: participants]
  United States | 46 | 45 | 47 | 138

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Incidence of Grade II-IV GVHD
Description: The primary outcome of this study is the cumulative incidence of grade II-IV acute GVHD up to Day 180 after stem cell infusion. Acute GHVD is graded according to the modified Glucksberg criteria (adapted from Thomas et al., NEJM ,1975, pp. 895-90), which is based on criteria by which the provider classifies acute GVHD per its objective organ staging. Acute GVHD is assessed in weekly standard of care visits post stem cell infusion and is captured in the protocol EDC upon evaluation of clinical notes up to Day 100. Data for acute GVHD organ staging and etiologies are collected in an acute GVHD separate case report form and do not include system organ class, expectedness or attribution.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A (Standard of Care) | Arm B (Experimental) | Arm C (Experimental)
Number analyzed (Participants) | 46 | 45 | 47
Percentage of participants | 33 [20 to 47] | 31 [18 to 45] | 21 [11 to 34]

2. Secondary Outcome: Percentage of Participants With Non-relapse Mortality
Description: Non-relapse mortality by 1 year after stem cell infusion.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A (Standard of Care) | Arm B (Experimental) | Arm C (Experimental)
Number analyzed (Participants) | 46 | 45 | 47
Percentage of participants | 11 [4 to 23] | 15 [6 to 28] | 6.5 [1.7 to 16]

3. Secondary Outcome: Percentage of Participants With Relapse
Description: Relapse relapse-cum-immunosuppression-free survival at 1 year after stem cell infusion
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A (Standard of Care) | Arm B (Experimental) | Arm C (Experimental)
Number analyzed (Participants) | 46 | 45 | 47
Percentage of participants | 24 [13 to 38] | 28 [15 to 42] | 36 [23 to 50]

4. Secondary Outcome: Percentage of Participants With Progression-free and Overall Survival
Description: Progression-free and overall survival 1 year post stem cell infusion
Time Frame: 1 year
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A (Standard of Care) | Arm B (Experimental) | Arm C (Experimental)
Number analyzed (Participants) | 46 | 45 | 47
Percentage of participants
  Progression free survival | 64 | 57 | 57
  Overall survival | 72 | 63 | 70

5. Secondary Outcome: Percentage of Participants With Chronic Graft Versus Host Disease
Description: Rates of chronic GVHD 1 year after stem cell infusion
Time Frame: 1 year
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A (Standard of Care) | Arm B (Experimental) | Arm C (Experimental)
Number analyzed (Participants) | 46 | 45 | 47
Percentage of participants | 59 | 55 | 55

ADVERSE EVENTS:
Time Frame: All adverse events experienced by participants will be collected from the time of the first dose of study treatment, through the study and until the final study visit. Participants continuing to experience toxicity at the off study visit may be contacted for additional assessments until the toxicity has resolved or is deemed irreversible.Participants will be followed for 1 year after transplantation or until death, whichever occurs first.
Description: AEs grade 3-5 & SAEs whether reported by the participant, discovered during questioning, directly observed, or detected by physical examination, laboratory test or other means, will be recorded in the participant's medical record and on the appropriate study-specific case report forms. Participants removed from study treatment for unacceptable AEs will be followed until resolution or stabilization of the AE. One participant was enrolled but immediately taken off study for alternative therapy.
Arm/Group | Arm A (Standard of Care) | Arm B (Experimental) | Arm C (Experimental)
Serious Adverse Events (participants affected / at risk) | 5/46 | 9/45 | 10/47
Other Adverse Events (participants affected / at risk) | 0/46 | 0/45 | 0/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Standard of Care) (N=46) | Arm B (Experimental) (N=45) | Arm C (Experimental) (N=47)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)
Treatment Related Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Malignant Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 4 (4)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Intracranial Hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus Bradycardia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalitis infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes